CLINICAL TRIAL: NCT02445820
Title: The Association Between Hydroxyethyl Starch 130/0.4 and Acute Kidney Injury After Cardiopulmonary Bypass: a Single-center Retrospective Study
Brief Title: HES and Acute Kidney Injury in Adult Cardiac Surgery
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Jean François Brichant, Professor of Anesthesia and Intensive Care Medicine, University of Liege
Other Study IDs: ANES2015002
Record Dates: First submitted 2015-05-05; First posted 2015-05-15 (Estimated); Last update posted 2015-10-30 (Estimated); Status verified 2015-10

CONDITIONS: Acute Kidney Injury After Adult Cardiac Surgery
MeSH Terms: interventions — Crystalloid Solutions; Plasmalyte A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- HES: Balanced HES 130/0.4 used as and pump prime and for intraoperative fluid therapy.
  Interventions: Drug: HES
- Crystalloid: Balanced Crystalloid used as a pump prime and for intraoperative fluid therapy.
  Interventions: Drug: Crystalloid

INTERVENTIONS:
Drug: HES — 2500 mL of balanced HES 130/0.4
  Other Names: Volulyte®
  Groups: HES
Drug: Crystalloid — 2500 mL of balanced crystalloid.
  Other Names: Plasmalyte A ®
  Groups: Crystalloid

SUMMARY:
This study retrospectively assess the effect or using balanced hydroxyethyl sctarch (HES) 130/0.4 or a balanced crystalloid solution as a pump prime and for intraoperative fluid therapy on the risk of early acute postoperative kidney injury in adult cardiac surgery patients.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 yo
* Having on pump cardiac surgery at CHU of Liège between April 2013 and June 2014

Exclusion Criteria:

* Off pump surgery
* Use of Blood or Albumin in the cardiopulmonary bypass priming solution
* Preoperative dialysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patients undergoing cardiac surgery
Sampling Method: Non-Probability Sample
Enrollment: 697 (Actual)
Dates: Start 2014-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
AKIN SCr | Forty eight hours
  Stage of acute kidney injury using the Acute Kidney Injury Network Classification omitting the diuresis criteria.

SECONDARY OUTCOMES:
AKIN SCr+UO | Forty eight hours
  Stage of acute kidney injury using the Acute Kidney Injury Network Classification including the diuresis criteria.
Postoperative dialysis | 30 days
  Requirement of postoperative renal replacement therapy
Respiratory complication | 30 days
  Need for reintubation, non-invasive ventilation or prolonged intensive care unit stay as a consequence of atelectasis, pulmonary edema or pneumonia.
ICU stay | 30 days
  Length of stay at the intensive care unit
Hospital stay | 30 days
  Length of stay at the hospital
30-day mortality | 30 days
  Death in hospital or within 30 days of surgery